CLINICAL TRIAL: NCT06280157
Title: A Long-term Follow-up Study to Assess the Persistence of Immunoglobin G (IgG) Antibodies to the GBS-NN/NN2 Vaccine After Vaccination With the GBS-NN/NN2 Vaccine in MVX0002 and/or in MVX0003
Brief Title: A Follow up Study of Group B Streptococcus (GBS)-NN/NN2 Vaccine in Healthy Volunteers
Status: Enrolling by invitation | Type: Observational
Sponsor: Minervax ApS (Other)
Collaborators: Simbec-Orion Group (Industry)
Responsible Party: Sponsor
Other Study IDs: MVX0007; 332126 (Other: IRAS)
Record Dates: First submitted 2024-02-19; First posted 2024-02-28 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Group B Streptococcus Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- One dose of GBS-NN/NN2: Participants who participated in study MVX003 and had received one dose of GBS-NN/NN2 prior to this study.
  Interventions: Biological: GBS-NN/NN2
- Two doses of GBS-NN/NN2: Participants who participated in study MVX002 and had received two doses of GBS-NN/NN2 prior to this study.
  Interventions: Biological: GBS-NN/NN2
- Three doses of GBS-NN/NN2: Participants who participated in study MVX002 and MVX003 and had received three doses of GBS-NN/NN2 prior to this study.
  Interventions: Biological: GBS-NN/NN2

INTERVENTIONS:
Biological: GBS-NN/NN2 — GBS-NN/NN2 containing 50 μg of GBS-NN and 50 μg of GBS/NN2

SUMMARY:
The goal of this follow-up study is to investigate the persistence of the immune response induced by the GBS-NN/NN2 vaccine in women who have participated in study MVX0002, and/or in study MVX0003 with GBS-NN/NN2 vaccine and received 1, 2 or 3 doses of GBS-NN/NN2. The main question it aims to answer is to determine the persistence of the immune response induced by the GBS-NN/NN2 vaccine by measuring antibody concentrations.

Participants who had received a primary course of GBS-NN/NN2 in Study MVX0002 and/or MVX0003 will be invited to return to have a single yearly blood sample of approximately 10 mL collected 2 to 5 years after the completion of the previous vaccination.

DETAILED DESCRIPTION:
This is a follow-up study to investigate the persistence of the immune response induced by the GBS-NN/NN2 vaccine. No vaccine or placebo will be administered. A single 10 mL blood sample will be collected from participants, every year, for a maximum of 4 years. Participants who had received a primary course of GBS-NN/NN2 in Study MVX0002 and/or MVX0003 will be invited to return to have a single yearly blood sample of approximately 10 mL collected 2 to 5 years after the completion of the previous vaccination.

Only participants that received two doses GBS-NN/NN2 in MVX0002 and all participants that received a single dose in MVX0003 will be eligible.

Hence, participants will have received:

One dose of GBS-NN/NN2 prior to this study, i.e., participants from MVX0003 who had not received GBS-NN/NN2 in MVX0002 and received a single dose in MVX0003.

Or two doses of GBS-NN/NN2 prior to this study, i.e., participants from MVX0002 who had received two doses of GBS-NN/NN2 in MVX0002 and did not take part in MVX0003.

Or three doses of GBS-NN/NN2 prior to this study, i.e., participants from MVX0003 who had received two doses of GBS-NN/NN2 in MVX0002 and received a single dose in MVX0003.

ELIGIBILITY:
Inclusion Criteria:

1. Women who have participated in study MVX0002, and/or in study MVX0003 with GBS-NN/NN2 vaccine and received 1, 2 or 3 doses of GBS-NN/NN2.
2. Able to voluntarily provide written informed consent to participate in the study.
3. Participant must be fit to participate in the study, as assessed by the investigator.
4. Participant must be able to comply with study procedures and provide at least 2 blood samples.

Exclusion Criteria:

1. Investigator site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the investigator, or MinervaX employees, including their family members.
2. Any known or suspected immunocompromising or immune suppressive condition (including conditions caused by certain immunocompromising/immunosuppressive medication), unless the condition is expected to normalise within 12 weeks after enrolment. If this is the case, then the subject can be enrolled but the blood sampling will be postponed until the condition has normalised.
3. Received systemic steroids in the 6 weeks before any blood sampling (inhaled and topical steroids are acceptable).
4. Received blood, blood products, plasma derivatives or any immunoglobulin preparations in the 12 weeks before any blood sampling.
5. While participants who are enrolled on this study will also be eligible for participation in other clinical trials which may be ongoing during the overall period of participation in this study, they are not allowed to participate in another vaccine study nor in a study involving a licensed or investigational drug which is known or suspected to have an impact on the immune response (immune compromising/suppressing/stimulating).

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: A minimum of 20 and a maximum of 55 female participants, all of whom received previous vaccination with GBS-NN/NN2 in the MVX0002 and MVX0003 studies, will be recruited.
Sampling Method: Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2024-01-18 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Antibody Concentration Specific for GBS-NN and GBS-NN2 | Baseline (Year 0), Years 1, 2, 3, 4
  Pharmacodynamic (PD) blood samples (10 mL) for antibody concentration specific for GBS-NN and GBS-NN2 will be collected during the study.
Ig G Antibody Responses Specific to Alpha like proteins (Alp): AlpCN | Baseline (Year 0), Years 1, 2, 3, 4
  Pharmacodynamic (PD) blood samples (10 mL) for antibody concentration specific for AlpCN, RibN, Alp1N and Alp2/3N will be collected during the study
Ig G Antibody Responses Specific to Alp: RibN | Baseline (Year 0), Years 1, 2, 3, 4
  Pharmacodynamic (PD) blood samples (10 mL) for antibody concentration specific for AlpCN, RibN, Alp1N and Alp2/3N will be collected during the study
Ig G Antibody Responses Specific to Alp: Alp1N | Baseline (Year 0), Years 1, 2, 3, 4
  Pharmacodynamic (PD) blood samples (10 mL) for antibody concentration specific for AlpCN, RibN, Alp1N and Alp2/3N will be collected during the study
Ig G Antibody Responses Specific to Alp: Alp2-3N | Baseline (Year 0), Years 1, 2, 3, 4
  Pharmacodynamic (PD) blood samples (10 mL) for antibody concentration specific for AlpCN, RibN, Alp1N and Alp2/3N will be collected during the study

CONTACTS AND LOCATIONS:
Overall Officials: Ebbe Englev, Study Director — Study Director
Locations (1):
- Simbec-Orion Clinical Pharmacology, Merthyr Tydfil, Pentrebach Merthyr Tydfil CF48 4DR, United Kingdom

IPD SHARING:
Plan to Share IPD: No